CLINICAL TRIAL: NCT02448888
Title: Prevention and Treatment of Chronic Low Back Pain Through an Adapted Exercise Program and General Exercise Recommendations Tailored to the Job on an Assembly Line Training Versus General Exercise Recommendations: Randomized Clinical Trial
Brief Title: Prevention and Treatment of Chronic Low Back Pain Through an Adapted Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: Mutua MAZ (Unknown); BSH electrodomésticos España S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTDLEF1
Record Dates: First submitted 2015-03-20; First posted 2015-05-20 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapted exercise (Experimental): The experimental group is going to follow a home-exercise program designed specifically to compensate the overloads and strength necessities of the workplace, the patient enter the description of the workplace in a mobile application and the APP shows the specific exercise that the patient needs to practice and general exercise recommendations.
  Interventions: Other: Adapted exercise
- General exercise recommendations (Experimental): The control group is going to receive general exercise recommendations (ACSM recommendations) with the same kind of APP to control the amount of exercise that each patient performs during the week.
  Interventions: Other: General exercise recommendations

INTERVENTIONS:
Other: Adapted exercise — 2 months, 3 times/week
  Arms: Adapted exercise
Other: General exercise recommendations — 2 months, 3 times/week
  Arms: General exercise recommendations

SUMMARY:
Objective: The purpose of this study is to investigate the effects of a adapted exercise program and general exercise recommendations compared with only general exercise recommendations for the management of chronic back pain among the workers of BSH (Bosch Siemens Hausgeräte), a manufacturing company.

DETAILED DESCRIPTION:
Design: Randomized controlled trial. Participants: Subjects (N_40 volunteers) experimental group (n_20) control group (n_20). All of the participants needs to be diagnosed with chronic back pain by a physician. Participants are going to be randomly assigned to two groups: a control group (CG), and experimental group (EG).

Intervention: The experimental group is going to follow a home-exercise program designed specifically to compensate the overloads and strength necessities of the workplace, the patient enter the description of the workplace in a mobile application (APP) and the APP shows specific exercises that the patient needs to practice. The exercise program includes muscle strengthening, flexibility, and endurance training, during 2 months, 3 times/week and generla recommendations. The control group is going to receive only general recommendation (ACSM recommendations) with the same kind of mobile application to control the amount of exercise that each patient performs during the week.

Data on pain intensity (BPI short form, Brief Pain Inventory), disability (Oswestry Low Back Pain Disability Questionnaire), functional assessment of the lumbar spine (EMG Flexion-relaxation test), amount of weekly physical activity (IPAQ), and number of sick leaves are going to be measured immediately before and after intervention and 3 months after the end of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* BSH industry workers.
* Spine pain diagnosed by a doctor, that has caused a previously sick-leave. The pain does not incapacitate to the patient to perform his job.
* In possession of a next-generation mobile.

Exclusion Criteria:

* Lumbar injury that does not let the patient performs his work or an exercise program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in lumbar pain intensity | Baseline, at the end of the two weeks training period and three months after the end of the training period.
  The assessment is performed with Brief Pain Index short form Self-administered questionnaire with 9 questions.
Change in disability caused by lumbar pain | Baseline, at the end of the two weeks training period and three months after the end of the training period.
  The assessment is performed with Oswestry Low Back Pain Disability Questionnaire,
Change in the functional assessment of the lumbar spine | Baseline, at the end of the two weeks training period and three months after the end of the train
  Functional assessment of the lumbar spine with EMG Flexion-relaxation test:

SECONDARY OUTCOMES:
Change in weekly physical activity amount | Baseline, at the end of the two weeks training period and three months after the end of the training period.
  Weekly physical activity performed by the patient assessed by the IPAQ
Incidence of sick-leave caused by lumbar pain | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Bataller, Study Director — San Jorge University; Cristina Cimarras, Principal Investigator — San Jorge University
Locations (2):
- Spain (2):
  - San Jorge University, Villanueva de Gállego, Zaragoza
  - BSH electrodomesticos España S.A, Zaragoza, Zaragoza